CLINICAL TRIAL: NCT02303132
Title: Ex Vivo Experiments to Evaluate the Role of Medication on the Colon Permeability in Microscopic Colitis
Brief Title: Ussing Experiments to Evaluate the Role of Medication-induced Microscopic Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL48505.068.14
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active MC (Other): Patients with active MC will be included
  Interventions: Other: Ussing experiment
- MC in remission (Other): Patients with MC in remission will be included
  Interventions: Other: Ussing experiment
- Controls (Other): Patients without MC will be included
  Interventions: Other: Ussing experiment

INTERVENTIONS:
Other: Ussing experiment — fresh colon mucosa (biopsy) of all participants will be mounted in an Ussing chamber and exposed to NSAIDs / PPI / control.

SUMMARY:
Medication use, especially NSAIDs and PPIs, prior to diagnosis is considered a risk factor for MC development. However, the exact pathophysiological mechanism is unclear. It is hypothesized that NSAIDs, PPIs, and SSRIs may have an effect on the colon permeability, due to an idiosyncratic reaction which results in a local immune response. MC patients are considered to be susceptible hosts, prone to react on administration of abovementioned drugs. In order to test this hypothesis and to generate new insights in the pathophysiology of MC, we want to perform an Ussing chamber experiment using fresh colon tissue samples. The primary objective is to assess ex vivo the effect of NSAIDs and PPIs on epithelial permeability of colon biopsy specimens of MC and non-MC patients, using the Ussing chamber system

ELIGIBILITY:
Inclusion Criteria:

* The indication for colonoscopy is a relapse of MC (active) / MC in remission (remission) / no MC (control)
* Patient is not treated with NSAIDs / PPI / SSRI in week before inclusion

Exclusion Criteria:

* Age below 18 years at the time of diagnosis
* Use of anticoagulants or immunosuppressive drugs
* Severe co-morbidities hindering an endoscopic procedure
* A previous history of any type of chronic colitis, IBS, IBD, colon carcinoma or (partial) colectomy
* A recent (last year) diagnosis of infectious diarrhea or radiation proctitis.
* Use of medication known to influence intestinal permeability
* Excessive alcohol usage (>20 standard units per week)
* Not capable of signing an informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Transepithelial electircal resistance | 2 hours

SECONDARY OUTCOMES:
Change in permeation of a fluorescent marker | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: A Masclee, PhD, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands